CLINICAL TRIAL: NCT03902054
Title: A Randomized, Blinded and Controlled Phase II Study to Evaluate the Safety and Immunogenicity of a Sabin Inactivated Poliovirus Vaccine (Vero Cell) in Infants.
Brief Title: Safety and Immunogenicity of a Sabin Inactivated Poliovirus Vaccine.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Beijing Minhai Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JSVCT042
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Polio and Post-Polio Syndrome
MeSH Terms: conditions — Postpoliomyelitis Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Experimental Group - High dosage (Experimental): Three intramuscular injections of the investigational vaccine(0.5 ml) on Day 0, Day 30 and Day 60 respectively; Intervention: Three-dose regimen of high dosage investigational sIPV
  Interventions: Biological: Three-dose regimen of high dosage investigational sIPV
- Experimental Group - Medium dosage (Experimental): Three intramuscular injections of the investigational vaccine(0.5 ml) on Day 0, Day 30 and Day 60 respectively; Intervention: Three-dose regimen of medium dosage investigational sIPV
  Interventions: Biological: Three-dose regimen of medium dosage investigational sIPV
- Experimental Group - Low dosage (Experimental): Three intramuscular injections of the investigational vaccine(0.5 ml) on Day 0, Day 30 and Day 60 respectively; Intervention: Three-dose regimen of low dosage investigational sIPV
  Interventions: Biological: Three-dose regimen of low dosage investigational sIPV
- Control Group -commercialized sIPV (Active Comparator): Three intramuscular injections of the investigational vaccine(0.5 ml) on Day 0, Day 30 and Day 60 respectively; Intervention: Three-dose regimen of commercialized sIPV
  Interventions: Biological: Three-dose regimen of commercialized sIPV
- Control Group -commercialized IPV (Active Comparator): Three intramuscular injections of the investigational vaccine(0.5 ml) on Day 0, Day 30 and Day 60 respectively; Intervention: Three-dose regimen of commercialized IPV
  Interventions: Biological: Three-dose regimen of commercialized IPV

INTERVENTIONS:
Biological: Three-dose regimen of high dosage investigational sIPV — The investigational vaccines were manufactured by Beijing Minhai Biotechnology Co. Ltd..
  Arms: Experimental Group - High dosage
Biological: Three-dose regimen of medium dosage investigational sIPV — The investigational vaccines were manufactured by Beijing Minhai Biotechnology Co. Ltd..
  Arms: Experimental Group - Medium dosage
Biological: Three-dose regimen of low dosage investigational sIPV — The investigational vaccines were manufactured by Beijing Minhai Biotechnology Co. Ltd..
  Arms: Experimental Group - Low dosage
Biological: Three-dose regimen of commercialized sIPV — The control vaccine was manufactured by Chinese Academy of Medical Sciences.
  Arms: Control Group -commercialized sIPV
Biological: Three-dose regimen of commercialized IPV — The control vaccine was manufactured by Sanofi Pasteur S.A (IMOVAX POLIO).
  Arms: Control Group -commercialized IPV

SUMMARY:
This study is a randomized, blinded and controlled phase II study to evaluate the safety and immunogenicity of a Sabin Inactivated Poliovirus Vaccine (sIPV) in Infants. A total of 600 infants aged 2 months (60~90 days) were randomized to receive five different vaccination regimens: three experimental groups (1, 2, and 3) received three doses of sIPV with high, medium, and low D antigen content, respectively, on the month 0,1,2 schedule; two control groups (4 and 5) received three doses of conventional IPV (cIPV, manufactured by Sanofi Pasteur) or sIPV (manufactured by the Institute of Medical Biology, the Chinese Academy of Medical Biology), respectively, on the same schedule. Serum samples were collected before the 1st dose and 30 days after the 3rd dose vaccination to assess the immunogenicity. Adverse events occurring within 30 days after each dose were collected to assess the safety.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer aged 2 months (60~90 days) old without prior vaccination of poliovirus and any contraindication for vaccination;
* Guardians of the participants should be capable of understanding the written consent form, and such form should be signed prior to enrolment;
* Complying with the requirement of the study protocol;
* Axillary temperature ≤ 37.0 °C;

Exclusion Criteria:

* Preterm or low birth weight infants;
* Congenital malformation, developmental disorders, genetic defects, or severe malnutrition;
* History of polio;
* Severe nervous system disease (epilepsy, seizures or convulsions) or mental illness;
* History of allergy to any vaccine, or any ingredient of the vaccine, or serious adverse reaction(s) to vaccination, such as urticaria, dyspnea, angioneurotic edema, abdominal pain, etc;
* Autoimmune disease or immunodeficiency/immunosuppressive;
* Bleeding disorder diagnosed by a doctor (e.g., coagulation factor deficiency, coagulation disorder, or platelet disorder) , or significant bruising or coagulopathy;
* Serious chronic diseases, respiratory diseases, cardiovascular diseases, liver or kidney diseases or skin diseases;
* Mother of the participant has HIV infection;
* Acute illness or acute exacerbation of chronic disease within the past 7 days;
* Had a high fever within the past 3 days (axillary temperature ≥ 38.0°C);
* Receipt of any subunit or inactivated vaccine within the past 7 day;
* Receipt of any live attenuated vaccine within the past 14 days;
* Receipt of any blood product within the past 3 months;
* Any other factor that, in the judgment of the investigator, suggesting the volunteer is unsuitable for this study;

Ages: 60 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2018-05-26 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
The seroconversion rates (SCRs) of each group after three-dose regimen | 28~42 days
  Subjects whose pre-immune antibody level < 1:8 and post-immune antibody level ≥ 1:8, or those whose pre-immune antibody level ≥ 1:8 and the increase of post-immune antibody level ≥ 4 folds are considered seroconverted.
The post-immune geometric mean titer (GMT) of each group after three-dose regimen | 28~42 days
  GMT of each group 28~42 days after three-dose regimen.
The geometric mean fold increase (GMI) of each group after three-dose regimen | 28~42 days
  The GMI is the increase of post-immune GMT from pre-immune GMT.

SECONDARY OUTCOMES:
The incidences of solicited adverse events (AEs) of each group | 7 days
  Solicited AEs occurred within 7 days after each injection will be collected.
The incidences of unsolicited adverse events (AEs) of each group | 30 days
  Unsolicited AEs occurred within 30 days after each injection will be collected.
The incidences of serious adverse events (SAEs) of each group | 30 days
  SAEs occurred within 30 days after each injection will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Jia S, Tang R, Li G, Hu Y, Liang Q. The effect of maternal poliovirus antibodies on the immune responses of infants to poliovirus vaccines. BMC Infect Dis. 2020 Aug 31;20(1):641. doi: 10.1186/s12879-020-05348-1. PMID 32867698